CLINICAL TRIAL: NCT01470911
Title: Phase-I Study in Healthy Male Subjects to Investigate Safety, Tolerability and Pharmacokinetics of Orally Inhaled Single Doses of SB010, a Human GATA-3-specific DNAzyme Solution for Nebulisation.
Brief Title: Safety, Tolerability, and Pharmacokinetics of Orally Inhaled DNAzyme Solution for Nebulisation in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sterna Biologicals GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SB010/01/2011; 2011-002916-10 (EudraCT Number)
Record Dates: First submitted 2011-10-31; First posted 2011-11-11 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: Antisense oligonucleotide; Asthma; Healthy subjects; Phase 1; Transcription factor GATA-3; Oral inhalation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SB010 (Experimental): The drug SB010 is administered in phosphate-buffered saline solution, inhaled via a controlled breathing system over a 5 to 10 min.
  Interventions: Drug: SB010
- Placebo (Placebo Comparator): The placebo (phosphate-buffered saline) is administered as a solution inhaled via a controlled breathing system over a 5 to 10 min.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB010 — Six ascending dose groups (DG) are planned, with a total of 48 subjects. DG 1 and 2 will consist of n=6 subjects (n=3 receiving SB010, n=3 placebo). The following DG will consist of n=9 subjects (n=6 receiving SB010, n=3 placebo). The number of subjects to be exposed to active compound will be limited on a particular study day. Subjects of a particular DG will be divided into subgroups and exposed to the drug on different days. In DG 1 and 2, the time interval between the two administrations of the first subgroup will be at least 2 hours. In DG 3-6, the time interval between two subsequent administrations will be at least 1 hour.
  Dose level (DL) 1: 0.4 mg hgd40/2 mL; DL 2: 2 mg hgd40/2 mL; DL 3: 5 mg hgd40/2 mL; DL 4: 10 mg hgd40/2 mL; DL 5: 20 mg hgd40/2 mL; DL 6: 40 mg hgd40/2 mL.
  Arms: SB010
Drug: Placebo — Six ascending dose groups (DG) are planned, with a total of 48 subjects. DG 1 and 2 will consist of n=6 subjects (n=3 receiving SB010, n=3 placebo). The following DG will consist of n=9 subjects (n=6 receiving SB010, n=3 placebo). The number of subjects to be exposed to active compound will be limited on a particular study day. Subjects of a particular DG will be divided into subgroups and exposed to the drug on different days. In DG 1 and 2, the time interval between the two administrations of the first subgroup will be at least 2 hours. In DG 3-6, the time interval between two subsequent administrations will be at least 1 hour.
  Arms: Placebo

SUMMARY:
Asthma is a chronic inflammatory bronchial disorder with three distinct components: airway hyper-responsiveness (respiratory hypersensitivity), airway inflammation, and intermittent airway obstruction. One of the characteristics of the disease is an inflammatory reaction of the immune system caused by cytokine production. A substantial number of asthma patients do not satisfactorily respond to steroid therapy and consequently have an unmet medical need for novel targeted therapies with improved specificity, tolerability, and compliance.

Novel therapeutic strategies for the treatment of chronic inflammatory diseases by targeting early disease-causing mechanisms are a promising approach for the treatment of asthma. The transcription factor GATA-3 plays a key role in mediating the asthmatic immune response and has been shown to be necessary and sufficient for the production of cytokines interleukin (IL)-4, IL-5, and IL-13. The active principle hgd40 of the investigational medicinal product SB010 belongs to a new class of antisense oligonucleotide therapeutics, the 10-23 DNA (deoxyribonucleic acid) zymes (antisense oligonucleotide). DNAzymes are catalytically active nucleic acids that cleave complementary RNA (ribonucleic acid) molecules. By cleaving GATA-3 mRNA hgd40 reduces specific cytokine production and thereby reduces key features of allergic airway inflammation.

DNAzymes are completely generated by chemical synthesis and can be produced under Good Manufacturing Practice (GMP) controlled conditions. The DNAzymes are not biological drugs, i.e. they are not generated by use of any living organism including cell culture or bacteria. The molecules are highly water-soluble and will be applied as solution directly in their synthesized form.

The current study will evaluate the safety and tolerability of increasing single doses of inhaled SB010 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participation in the trial prior to trial start and any trial-related procedure.
* Healthy male Caucasian subject - healthy based on a screening examination including medical history, without clinically relevant pathologies, physical examination, vital signs, ECG assessment, pulmonary function testing, and clinical laboratory results.
* Body weight according to a body mass index (BMI) between 18 and 29 kg/m2 (inclusive); body weight between 60 and 90 kg.
* Non-smokers or ex-smokers (stopped smoking for at least 5 years prior to start of the clinical study).
* Ability to inhale in an appropriate manner.

Exclusion Criteria:

* History or current evidence of clinically relevant allergies or idiosyncrasy to any drug or food.
* History of allergic reactions to any active or inactive component of the study medication.
* History or current evidence of any clinically relevant pulmonary, cardiovascular, hepatic, renal, gastrointestinal, haematological, endocrinological, metabolic, neurological, or psychiatric disease within the last 2 years.
* ECG abnormalities of clinical relevance (e.g., QTc according to Bazett's ³440 ms, PR ³210 ms; or QRS ³120 ms).
* Subjects with a resting heart rate <50 bpm, systolic blood pressure <100 mmHg, diastolic blood pressure <60 mmHg.
* Proneness to orthostatic dysregulation, fainting, or blackouts.
* History or presence of any malignancy except for basalioma.
* Abnormalities in clinical chemical or haematologic variables considered medically relevant by the investigator.
* Chronic or acute infections.
* Positive results in any of the following virology tests: human immunodeficiency virus (HIV) antibodies and antigen, Anti-hepatitis B-core antibody, hepatitis B surface antigen (HBsAg) and anti-hepatitis C virus antibody.
* Positive drug screen.
* History of previous administration of any registered or investigational oligonucleotide-based drug.
* History or presence of alcohol or drug abuse.
* Treatment with any known enzyme inducing or inhibiting agents (e.g., St. John's Wort (Johanniskraut), barbiturates, phenothiazines, cimetidine, ketoconazole, etc.) within 30 days before administration of IMP or during the trial.
* Use of any medication (including over-the-counter medication, herbal products) except allowed concomitant medication within 2 weeks (for biologics: 6 months) before administration of IMP or within <10 times the elimination half-life of the respective drug, or the duration of the pharmacodynamic effect, whatever is longer.
* Consumption of any enzyme inducing or inhibiting aliments and beverages (e.g., broccoli, Brussels sprout, grapefruit, grapefruit juice, star fruit etc.) within 14 days prior to the IMP administration or during the trial.
* Consumption of any caffeine- or theophylline-containing product 48 h before administration of IMP.
* Consumption of alcohol within 48 h before administration of IMP.
* Vegetarian diet or other dietary habits, which would preclude the subject's acceptance of standardised meals.
* Surgery of the gastrointestinal tract except for appendectomy or herniotomy.
* Planned donation of germ cells, blood, organs, bone marrow during the course of the trial or within 6 months thereafter.
* Participation in another clinical trial with an investigational drug or device within the last 3 months. For biologics, the minimum exclusion period is at least 6 months or the time of duration of the pharmacodynamic effect or 10 times the half-life of the respective drug whatever is longer before inclusion in this trial.
* Blood donation within the last 30 days before screening.
* Lack of ability or willingness to give informed consent.
* Anticipated non-availability for trial visits/procedures.
* Anticipated lack of willingness or inability to cooperate adequately.
* Vulnerable subjects (e.g., persons kept in detention).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Limiting dose of inhaled ascending single dose of SB010. | Study period 4 days, follow up visit 12±2 days, end of study day 60±4 days; maximum of 78 days for a particular subject.
  Safety will be monitored as adverse events, vital signs, clinical chemistry, haematology, urinalysis, electrocardiogram, pulmonary function testing, body temperature, overall tolerability.

SECONDARY OUTCOMES:
Number of participants with any dose-limiting adverse effects. | Study period 4 days, follow up visit 12±2 days, end of study day 60±4 days; maximum of 78 days for a particular subject.
  Safety will be monitored as adverse events, vital signs, clinical chemistry, haematology, urinalysis, electrocardiogram, pulmonary function testing, body temperature, overall tolerability.
Maximum tolerated dose. | Study period 4 days, follow up visit 12±2 days, end of study day 60±4 days; maximum of 78 days for a particular subject.
  Safety will be monitored as adverse events, vital signs, clinical chemistry, haematology, urinalysis, electrocardiogram, pulmonary function testing, body temperature, overall tolerability.
Single-dose plasma concentration of hgd40 over time after inhalation of SB010. | Day 1 to 4 of the study.
  The following pharmacokinetic parameters will be determined in plasma samples over 4 days: Area under the plasma concentration-time curve; Concentration maximum; Time of maximum concentration; Apparent terminal elimination half-life; Area under the concentration-time curve until the last sampling time;
Feasibility of the inhalative technique. | Day 1.
  Study participants will be instructed on the correct inhalation technique. Ability to breath in through the mouth and exhale through the nose will be assessed during the inhalation procedure. Forced Expiratory Volume in 1 second(FEV1*) will be monitored at screening and throughout the study after the single dose of the study drug: Days 1, 2, 3, 4, 12±2, and 60±4
  *FEV1 = the maximal amount of air forcefully exhaled in one second

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Timmer, MD, Principal Investigator — CRS-Mannheim GmbH, Germany
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany